CLINICAL TRIAL: NCT02113293
Title: A Phase 1, Two Period, Double-blind, Randomised, Placebo-controlled, Cross- Over Study Investigating the Safety, Local Tolerability and Systemic Exposure of Cyclosporine A and Placebo (Vehicle) Following Single and Multiple Ocular Doses of CyclASol® and Placebo in Healthy Volunteers (CYS-001).
Brief Title: CyclASol® Phase 1 Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novaliq GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYS-001; 2013-005423-16 (EudraCT Number)
Record Dates: First submitted 2014-04-07; First posted 2014-04-14 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: phase I study; tolerability; safety; CyclASol®; eye drops

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CyclASol® (Experimental): CyclASol®
  Interventions: Drug: CyclASol®
- Placebo (Placebo Comparator): Placebo (vehicle)
  Interventions: Drug: Placebo (vehicle)

INTERVENTIONS:
Drug: CyclASol® — Cyclosporine A Solution
  Arms: CyclASol®
Drug: Placebo (vehicle) — Vehicle Solution
  Arms: Placebo

SUMMARY:
This study is intended to investigate the tolerability and the safety of Cyclosporine A containing CyclASol® eye drops compared to Placebo (vehicle) in a cohort of healthy volunteers. Subjects will be randomly assigned to dosing with CyclASol® eye drops or Placebo (vehicle) in the first part (first period) of the study, and switched to the alternative dosing in the second part (second period) of the study. An ophthalmological assessment of the eyes will be performed, and a questionnaire will be issued in the beginning and after each dosing. Additionally physical examinations, safety laboratory and ECGs will be performed, and blood samples will be analyzed for Cyclosporine A and Placebo (vehicle).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subject aged 18 - 45 years
* Nonsmoker, for at least three months prior to first dose of trial medication
* BMI from 18.5 to 29.9 (kg/m2)
* Corneal/Conjunctival staining Oxford grading = 0°
* Schirmer I more than 10 mm/5min
* Tear Film Break-Up Time (TFBUT) equal or more than 10 s
* Intra-ocular pressure between 10 and 20 mmHg
* Normal funduscopy
* Subject will have given their voluntary written informed consent to participate in the study in their own language and are willing to comply with the protocol

Exclusion Criteria:

* History of clinically relevant allergy (except for untreated, asymptomatic, seasonal allergies at time of dosing)
* History of dry eye disease, ocular surgery, corneal disease
* Known hypersensitivity to the drug substance
* Limbal stem cell deficiency
* Cicatricial pemphigoid
* Glaucoma or known steroid response on intraocular pressure
* Ocular allergy or incompatibility against Ciclosporin or semifluorinated alkanes
* Punctual occlusion
* Corrected vision with glasses less than 0.7 on one or both eyes
* Contact lens wear 3 weeks before to the planned first drug administration and/or during the study
* Acute infection of ocular surface (bacterial, viral, fungal...)
* Acute trauma of ocular surface
* No acceptable methods of birth control
* Pregnancy or breast-feeding period (females only)
* Use of any drugs whatsoever (including vitamins and herbals) for fourteen (14) days prior to the planned first drug administration (excluding contraceptives in women and single use of paracetamol or ibuprofen)
* Topical or systemic therapy with steroids, Ciclosporin, non-steroidal anti- inflammatory drugs, tetracyclines or other immunomodulatory substances within last 90 days prior to the planned first drug administration or during this trial

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Local tolerability measured by the rate and severity of drug-related adverse events of the eyes | 45 days
  Multiple ophthalmologic assessments are performed in order to determine adverse effects of the investigational medicinal product on structures of the eye and its physiology.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Beckert, MD, Study Director — Novaliq GmbH
Locations (1):
- Neu-Ulm, Germany